CLINICAL TRIAL: NCT07386327
Title: The Effect of Diluting Bupivacaine With 5% Dextrose and 0.9% NaCl on Block Success and Duration of Analgesia in Infraclavicular Block
Brief Title: Impact of Bupivacaine Dilution With Dextrose or Saline on Infraclavicular Block Outcomes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Burçin Alaçam, MD (Other)
Responsible Party: Sponsor-Investigator, Burçin Alaçam, MD, Anesthesiology Specialist, Sakarya University
Organization: Sakarya University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SAU-ANE-BA-03
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Infraclavicular Brachial Plexus Block; Dextrose; Bupivacaine; Block Success; Postoperative Analgesia
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups. In the first group, bupivacaine will be diluted with 5% dextrose in water (D5W), and in the second group, bupivacaine will be diluted with 0.9% sodium chloride (normal saline). All patients will undergo ultrasound-guided infraclavicular brachial plexus block using the assigned study solution. Block success, duration of analgesia, and secondary block characteristics will be compared between the two groups.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The anesthesiologist performing the block will be aware of the study solution due to preparation requirements. Patients, outcome assessors, and data analysts will be blinded to group allocation to minimize assessment and analysis bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group D (Experimental): Participants in this group will receive an ultrasound-guided infraclavicular brachial plexus block using bupivacaine diluted in a 1:1 ratio with 5% dextrose in water (D5W) to achieve a predetermined total injection volume (e.g., total volume of 30 mL). The block will be performed under standardized aseptic conditions by an experienced anesthesiologist. Block success, sensory and motor block characteristics, duration of analgesia, and postoperative analgesic requirements will be assessed and recorded.
  Interventions: Diagnostic Test: Blocked and analgesia time
- Group S (Experimental): Participants in this group will receive an ultrasound-guided infraclavicular brachial plexus block using bupivacaine diluted in a 1:1 ratio with 0.9% sodium chloride (normal saline) to achieve a predetermined total injection volume (e.g., total volume of 30 mL). The block will be performed under standardized aseptic conditions by an experienced anesthesiologist. Block success, sensory and motor block characteristics, duration of analgesia, and postoperative analgesic requirements will be assessed and recorded.
  Interventions: Diagnostic Test: Blocked and analgesia time

INTERVENTIONS:
Diagnostic Test: Blocked and analgesia time — All eligible participants will be informed in detail about the study objectives, procedures, potential risks, and benefits by the responsible investigator, and all questions will be answered prior to enrollment. Written informed consent will be obtained from each participant before any study-related procedures are initiated.
  Following the ultrasound-guided infraclavicular block, sensory block assessment will be performed using a sterile single-use needle for a pinprick test. Light punctate stimuli will be applied to dermatomal areas corresponding to the branches of the brachial plexus on the blocked extremity. Participants will be asked to compare the sensation with the contralateral limb and to report the perceived sensation as "normal," "reduced," or "absent." Sensory block assessments will be performed at 5, 10, 15, 20, and 30 minutes after block administration. Sensory block onset time will be defined as the time point at which the participant reports absence of pinprick sensation

SUMMARY:
D5W) has long been used as an intravenous fluid for hydration and energy supplementation and has recently gained increasing clinical interest in perineural injection therapies and ultrasound-guided hydrodissection. D5W has been shown to improve pain and functional outcomes in entrapment neuropathies by mechanically releasing perineural adhesions and potentially modulating neurogenic inflammation. In contrast, 0.9% sodium chloride (normal saline) is routinely used as a dilution medium for local anesthetics in peripheral nerve blocks; however, emerging evidence suggests that alternative diluents such as D5W may influence block onset and efficacy.

The infraclavicular block is a commonly used ultrasound-guided technique for brachial plexus anesthesia, providing reliable anesthesia and postoperative analgesia for upper extremity surgery. This study aims to compare the effects of diluting bupivacaine with either D5W or 0.9% NaCl on block success and duration of analgesia in patients undergoing infraclavicular block. Secondary outcomes include block onset characteristics, sensory and motor block profiles, and perioperative analgesic requirements. The findings may help determine whether D5W represents a safe and effective alternative diluent to saline in routine regional anesthesia practice.

DETAILED DESCRIPTION:
D5W) has traditionally been used as an intravenous fluid to provide hydration and caloric support. In recent years, D5W has gained increasing attention for its use in innovative perineural injection therapies and ultrasound-guided hydrodissection techniques, particularly in the management of peripheral nerve entrapment syndromes. Clinical and randomized controlled studies have demonstrated that perineural D5W hydrodissection can mechanically separate fibrotic tissues surrounding compressed nerves, improve perineural blood flow, reduce pain, and enhance sensory and functional recovery in conditions such as carpal tunnel syndrome and meralgia paresthetica. Beyond its mechanical effects, D5W is also thought to modulate neurogenic inflammation, regulate nociceptive C-fiber activity through local glucose-related mechanisms, and potentially promote neuroregenerative processes.

In routine regional anesthesia practice, 0.9% sodium chloride (normal saline) is the most commonly used diluent for local anesthetics to achieve the desired volume and concentration for peripheral nerve blocks. However, experimental and clinical data suggest that the sodium content and physicochemical properties of saline may influence the onset and quality of neural blockade. Some studies have reported earlier sensory block onset when local anesthetics are diluted with D5W rather than saline, suggesting that the choice of diluent may affect block characteristics.

The infraclavicular brachial plexus block is a well-established ultrasound-guided technique that provides reliable anesthesia and postoperative analgesia for surgeries involving the mid and distal upper extremity. Visualization of neural structures allows optimized local anesthetic spread and consistent block performance in routine clinical practice.

This study is designed to evaluate the effect of diluting bupivacaine with either D5W or 0.9% NaCl on block success and duration of analgesia in patients undergoing ultrasound-guided infraclavicular block. Secondary outcomes will include onset time of sensory and motor block, block quality, postoperative analgesic consumption, and safety parameters. By investigating an alternative dilution strategy, this study aims to contribute to optimizing peripheral nerve block techniques and improving patient-centered clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree to participate in the study and provide written informed consent
* Patients scheduled for elective upper extremity surgery for whom infraclavicular block is considered appropriate for anesthetic management
* Age between 18 and 65 years
* American Society of Anesthesiologists (ASA) physical status I-III
* Patients with a normal neurological examination in the extremity scheduled for peripheral nerve block

Exclusion Criteria:

* Patients who decline to participate in the study or refuse to provide informed consent
* History of allergy or hypersensitivity to study medications
* Body mass index (BMI) ≥ 30 kg/m²
* Body weight less than 40 kg
* Age below 18 years or above 65 years
* History of significant cardiac disease (e.g., arrhythmia, conduction disorders)
* Presence of coagulopathy (international normalized ratio [INR] > 1.5 and/or platelet count < 100,000/mm³)
* Hepatic failure or significant liver dysfunction
* Pregnant patients
* Infection at the planned peripheral block site
* Presence of neurological deficit in the extremity planned for peripheral nerve block
* Patients with uncontrolled diabetes mellitus and/or established diabetic neuropathy
* American Society of Anesthesiologists (ASA) physical status IV

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Sensory block onset time | Assessed at 5, 10, 15, 20, and 30 minutes after block administration.
  Sensory block onset time will be defined as the time from completion of the ultrasound-guided infraclavicular block until the participant reports complete loss of pinprick sensation in the dermatomal areas corresponding to the branches of the brachial plexus, assessed using a sterile pinprick test.

SECONDARY OUTCOMES:
Motor block duration | From block performance until complete motor recovery (up to 24 hours postoperatively).
  Motor block duration will be defined as the time from onset of motor block (Modified Upper Extremity Bromage Scale ≥1) until full recovery to Bromage score 0.
Intraoperative need for additional anesthetic or analgesic intervention | During the intraoperative period.
  Requirement for supplemental anesthetic or analgesic interventions during surgery will be recorded as a binary outcome (yes/no) and as total additional drug consumption if applicable.
Postoperative analgesic efficacy | Postoperative 2, 6, 12, and 24 hours.
  Postoperative pain intensity will be assessed using the Visual Analog Scale (VAS; 0 = no pain, 10 = worst imaginable pain) at postoperative 2, 6, 12, and 24 hours.

IPD SHARING:
Plan to Share IPD: No